CLINICAL TRIAL: NCT05039580
Title: A Clinical Trial of PD-1 Monoclonal Antibody as First-line Induction Therapy for EBV-associated Hemophagocytic Syndrome (EBV-HLH) or Chronic Active EBV Infection (CAEBV)
Brief Title: Programmed Cell Death Protein-1 (PD-1) Monoclonal Antibody for EBV-HLH and CAEBV as First-line Therapy
Acronym: SEHC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBV and CAEBV 001
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-07

CONDITIONS: EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — spartalizumab; ruxolitinib; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 monoclonal antibody group (Experimental): PD-1 monoclonal antibody 200mg is infused intravenously once for patients whose age >=18 years, or age <18 years but weight >=40kg. While for patients age <18 years, the dose of PD-1 monoclonal antibody is 3mg/kg.
  Interventions: Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: PD-1 monoclonal antibody — PD-1 monoclonal antibody is a new attempt treatment, and ruxolitinib and/or low-dose dexamethasone can reduce the inflammation that occur in EBV-HLH or CAEBV.
  Other Names: ruxolitinib; dexamethasone

SUMMARY:
EBV-HLH and CAEBV are both caused by EBV infection, part of them can rapidly lead to a syndrome of severe, life-threatening hyper-inflammation, with poor prognosis. Currently, the most effective treatment remains unknown. This study is trying to evaluate the efficacy and safety of PD-1 monoclonal antibody as a first-line therapy for EBV-HLH and CAEBV.

DETAILED DESCRIPTION:
Eligible patients who were diagnosed with EBV-HLH or CAEBV, age between 12 and 70 years, were enrolled in this study. All of them need to sign the informed consent first.

PD-1 monoclonal antibody 200mg is infused intravenously once for patients whose age >=18 years, or age <18 years but weight >=40kg. While for patients age <18 years, the dose of PD-1 monoclonal antibody is 3mg/kg. Besides, optimal supportive care is necessary.

Ruxolitinib and/or low-dose glucocorticoid can be used to reduce inflammation.

Cerebrospinal fluid parameters are examined, and methotrexate 15mg combined with dexamethasone will be intrathecal injected without contraindications.

Clinical and laboratory indicators are investigated weekly to evaluate the efficacy and toxicity.

If patients achieve partial response/complete response within 14 days after PD-1 monoclonal antibody, the clinical observations are stopped. If not, the observation period is prolonged to 21 days.

If disease progress at day 21, this study is terminated, and the patient should be transfer to other treatments as soon as quickly.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of EBV-HLH or CAEBV.
2. Newly diagnosed patients.
3. Eastern Cooperative Oncology Group score 0-3.
4. Total bilirubin <= 10 times of upper limit of normal (except for those caused by EBV-HLH or CAEBV), and serum creatinine <= 1.5 times of upper limit of normal.
5. Serum HIV antigen or antibody is negative.
6. Hepatitis C virus (HCV) antibody is negative, or HCV antibody is positive, but HCV-RNA is negative.
7. Both HbsAg and HbcAb for Hepatitis B virus (HBV) are negative. If not, the quantification of HBV-DNA needs to be <1*10e3 IU/ml.
8. The patient or his/her guardian must be able to understand and be willing to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. Non EBV-HLH or CAEBV patients.
2. Refractory or relapsed EBV-HLH or CAEBV.
3. Heart function above grade II (NYHA).
4. Patients suffered from other uncontrollable active infections.
5. Pregnant or lactating women.
6. Patients with mental disorders and cannot cooperate with the requirements of research, treatment and monitoring.
7. Active visceral bleeding.
8. Allergic to PD-1 monoclonal antibody.
9. Patients with known autoimmune diseases.
10. Participate in other clinical research at the same time.
11. The investigator judges that the patient has other reasons not suitable for this study, or participating in the study will bring great risks to the patient.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 weeks
  complete response and/or partial response rate
EBV-DNA viral load | 3 weeks
  EBV-DNA copy by polymerase chain reaction

SECONDARY OUTCOMES:
Time for treatment works | 3 weeks
  Time to achieve partial response or complete response
Toxicity of PD-1 monoclonal antibody | 3 weeks
  Side effects related to immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No